CLINICAL TRIAL: NCT01119677
Title: A Randomized, Three-Arm, Dose-Blinded, Parallel-Group Study to Determine the Effect of Avonex® Dose Titration on the Severity and Incidence of Interferon Beta-1a-Related Flu Like Symptoms in Healthy Volunteers
Brief Title: A Study of Avonex to Determine the Effects of Dose Titration on the Incidence of Flu Like Symptoms in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 108HV103
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): No dose titration
  Interventions: Drug: Avonex
- Group 2 (Experimental): Fast dose titration
  Interventions: Drug: Avonex
- Group 3 (Experimental): Slow dose titration
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: Avonex — Group 1 subjects will receive weekly Avonex 30 mcg (full dose) IM injections from Week 1 to Week 8. Group 2 subjects will titrate in quarter dose increments every week up to a full dose of Avonex over a 3 week period from Week 1 to Week 3 and then continue on full dose from Week 4 to Week 8. Group 3 subjects will titrate in quarter dose increments every 2 weeks up to a full dose of Avonex over a 6 week period from Week 1 to Week 6 and continue on full dose from Week 7 to Week 8

SUMMARY:
The primary objective of the study is to determine whether titration of Avonex reduces the severity of flu-like symptoms (FLS). Secondary objectives of this study are to determine whether titration of Avonex reduces the incidence of FLS and to evaluate the overall safety and tolerability of Avonex intramuscular (IM) injections.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a Body Mass Index of 19 to 30 kg/m2, and a minimum body weight of 50.0 kg at Screening.
* Female participants of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Key Exclusion Criteria:

* Known history of or positive test result for human immunodeficiency virus (HIV), hepatitis C virus (test for hepatitis C virus antibody [HCV Ab]) or hepatitis B virus (test for hepatitis B surface antigen [HBsAg] and hepatitis B core antibody [HBcAb])
* Known history of chronic fatigue syndrome or fibromyalgia
* Within one month, flu-like illnesses (e.g., gastroenteritis, upper respiratory infection, common cold)
* History of severe allergic reactions to any drug or anaphylactic reactions
* Known allergy to Avonex or any of its components
* Serious infection (e.g., pneumonia, septicemia) within the 3 months prior to Screening or active bacterial or viral infection
* History of alcohol or substance abuse (as defined by the Investigator)
* Female participants who are pregnant or currently breastfeeding
* Any previous treatment with any interferon product.10. Vaccinations within 2 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Blood donation within 30 days prior to Screening
* Use of any tobacco product more than 5 times within 30 days prior to Screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05-05 (Actual); Primary Completion 2010-10-23 (Actual); Study Completion 2010-10-23 (Actual)

PRIMARY OUTCOMES:
To determine whether titration of Avonex reduces the incidence of flu like symptoms | 8 weeks

SECONDARY OUTCOMES:
To evaluate the overall safety and tolerability of Avonex IM injections | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Matson MA, Zimmerman TR Jr, Tuccillo D, Tang Y, Deykin A. Dose titration of intramuscular interferon beta-1a reduces the severity and incidence of flu-like symptoms during treatment initiation. Curr Med Res Opin. 2011 Dec;27(12):2271-8. doi: 10.1185/03007995.2011.630720. Epub 2011 Oct 28. PMID 21988668